CLINICAL TRIAL: NCT02518893
Title: Health Research Participation: Experiences and Decisions of Military Members
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: TriService Nursing Research Program (Other); Madigan Army Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wendy Cook, PhD, School of Nursing, University of Washington
Other Study IDs: 48058; HU0001-14-1-TS07 (N14-P10) (Other Grant/Funding Number: TriService Nursing Research Program); IRB #215029 (Other: Madigan Army Medical Center)
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Decision Making; Life Experiences
Keywords: Military Personnel; Air Force Personnel; Army Personnel; Navy Personnel; Armed Forces Personnel; Marines; Soldiers; Sailors; Airmen; Decision Making; Research Subjects; Life Experiences; Patient Participation; Refusal to Participate; Healthcare Research; Qualitative Research; Interview; Interviews, Telephone; Ethics, Research
MeSH Terms: conditions — Patient Participation | interventions — Demography; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Demographic Data — Demographic data will be collected from up to 50 service members who have participated in health research or who have previously declined research participation.
Other: Interview — Up to 40 service members will participate in individual, in-depth, semi-structured interviews in person or via telephone.

SUMMARY:
The purpose of the study is to describe service members' experiences as participants in health research, including their reasons for deciding for or against research participation.

DETAILED DESCRIPTION:
Recent studies of war injuries have included as research participants US military service members returning from wars in Iraq and Afghanistan. Despite the increased demand for military relevant research, little is known about the recent experiences of service members as research participants or about their research participation decisions.

The study aims are to: 1). Describe the experiences of military service members who have participated in health research; 2). Explore the reasons military service members decide for or against participation in health research; and 3). Identify effective strategies for promoting military service members' participation in research.

Demographic data will be collected from up to 50 service members who have participated in health research or who have previously declined research participation.

Up to 40 service members will participate in individual, in-depth, semi-structured interviews in person or via telephone.

ELIGIBILITY:
Inclusion Criteria:

* current US military member of any branch of service at time of screening
* experience as a research participant and/or previously declined participation in at least one health research study within the past three years
* age 18-80 years
* willing to participate in this study
* willing to be interviewed
* consents to participate

Exclusion Criteria:

* people who do not meet inclusion criteria
* unable to verbally communicate in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current United States military service members (active duty, reserve, or guard) of any service branch who have participated in military or civilian health care research within the past three years or who have declined research participation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Experiences of health research participation | Within past three years
  Self-reports of health research participation experiences
Research participation decisions | Within past three years
  Self-reports of research participation decisions

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A Cook, PhD, MA, RN, Principal Investigator — University of Washington
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Background] Cook WA, Doorenbos AZ. Indications of Recruitment Challenges in Research with U.S. Military Service Members: A ClinicalTrials.gov Review. Mil Med. 2017 Mar;182(3):e1580-e1587. doi: 10.7205/MILMED-D-16-00225. PMID 28290928
- [Background] Cook WA, Doorenbos AZ, Bridges EJ. Trends in Research with U.S. Military Service Member Participants: A Population-Specific ClinicalTrials.gov Review. Contemp Clin Trials Commun. 2016 Aug 15;3:122-130. doi: 10.1016/j.conctc.2016.04.006. Epub 2016 Apr 30. PMID 27822569
- [Result] Cook WA, Melvin KC, Doorenbos AZ. US Military Service Members' Reasons for Deciding to Participate in Health Research. Res Nurs Health. 2017 Jun;40(3):263-272. doi: 10.1002/nur.21785. Epub 2017 Feb 10. PMID 28185285